CLINICAL TRIAL: NCT05355272
Title: Growth Hormone Replacement Therapy in Veterans With Gulf War Illness and Adult Growth Hormone Deficiency
Brief Title: Growth Hormone Replacement in Veterans With GWI and AGHD (GWIT)
Acronym: GWIT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ricardo Jorge, MD, Professor of Psychiatry and Behavioral Sciences, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-49490; CDMRP-GW200072 (Other: CDMRP)
Record Dates: First submitted 2022-04-20; First posted 2022-05-02 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Gulf War Syndrome; Adult Growth Hormone Deficiency
Keywords: recombinant human growth hormone; growth hormone replacement therapy
MeSH Terms: conditions — Persian Gulf Syndrome; Dwarfism, Pituitary | interventions — Growth Hormone; Human Growth Hormone

STUDY DESIGN:
Intervention Model Description: This is a single-arm futility trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Growth Hormone Replacement Therapy (Experimental): Patients will be started at a dose of 200-300 mcg/d of daily injections of GHRT. A biweekly titration period of 6 weeks will be performed in increments of 100 mcg/d as needed until IGF-1 levels are between +1 and +2 standard deviation score, up to a maximum dose of 2,000 mcg/d, provided the dose is well tolerated.
  The duration of the intervention is 6-months. Participants will complete in-clinic follow-up visits at Days 14, 40, 65, 90, and 180. The primary outcome will be the change in truncal fat mass percentage from baseline to six months measured by dual-energy x-ray absorptiometry (DEXA).
  Interventions: Drug: Recombinant human growth hormone

INTERVENTIONS:
Drug: Recombinant human growth hormone — recombinant human growth hormone (rhGH)
  Other Names: Somatropin; Genotropin; Humatrope; Norditropin

SUMMARY:
The goal of the GWIT Study is to assess whether growth hormone replacement therapy is a safe and effective treatment for veterans with Gulf War Illness (GWI) and adult growth hormone deficiency (AGHD). The main questions the study aims to answer are:

1. Is growth hormone effective at reducing fat in the trunk of the body and symptoms of GWI among veterans with GWI and growth hormone deficiency?
2. Do the results of the study suggest there is merit in pursuing a larger trial to examine the efficacy of growth hormone as a treatment for growth hormone deficiency among veterans with Gulf War Illness?

To determine eligibility for the study, veterans will be asked to complete several assessments including questionnaires, blood tests, and a scan of the brain. Participants who qualify for the study will receive recombinant human growth hormone for 6-months. A body composition scan will be performed at Day1, Day 90, and Day 180 of the intervention. Questionnaires and cognitive tests will also be collected before and after the trial.

DETAILED DESCRIPTION:
Veterans with Gulf War Illness (GWI) often experience a range of debilitating symptoms, including fatigue, chronic pain, depression, anxiety, and cognitive dysfunction. The factors contributing to these symptoms remain poorly understood, but adults with adult growth hormone deficiency (AGHD) experience similar symptoms. Growth hormone replacement therapy has been shown to improve fatigue, chronic pain, mood, cognitive function, and quality of life. Approximately 1 in 3 Veterans diagnosed with GWI also tests positive for AGHD, raising the question of whether growth hormone replacement therapy (GHRT) could be a potential avenue for improving their quality of life.

The objective of this research is to conduct a clinical trial to determine whether GHRT can improve body composition, cognitive function, sleep quality, fatigue, and mood in Veterans with GWI and AGHD. Data from this study will also provide important information on the safety of the intervention.

This research has the potential to reshape our understanding of GWI and its therapeutic management. If GHRT proves efficacious, it could prompt widespread screening and treatment for growth hormone deficiency among Gulf War Veterans, potentially ameliorating their symptoms and enhancing their functional recovery. Furthermore, the findings of this study may influence clinical practice guidelines, facilitating more effective communication and collaboration among Veterans, caregivers, researchers, and healthcare providers.

ELIGIBILITY:
Inclusion Criteria:

1. veteran of the Gulf War conflict with a history of deployment to Operation Desert Storm or Desert Shield between 1990-91
2. age less than or equal to 64 years old
3. have a diagnosis of Gulf War Illness assessed by study investigators
4. have adult growth hormone deficiency diagnosed by glucagon stimulation test (cut point 3.0 mcg/L if BMI is less than or equal to 25 or 1.0 mcg/L if BMI is greater than 25)
5. 4-week stability on any psychotropic medications
6. 3-month stability on all hormone treatments
7. able and willing to provide informed consent to participant in the study and complete study protocol

Exclusion Criteria:

1. history of a psychiatric disorder with substantial impact on functional status or quality of life (e.g., schizophrenia, schizoaffective disorder, bipolar, or other psychotic disorder)
2. history of neurologic disorder other than traumatic brain injury with substantial impact on the quality of life
3. other known cause for growth hormone deficiency (GHD) including history of childhood onset GHD, hypothalamic/pituitary disease, history of brain radiation, or genetic mutations known to lead to GHD
4. active suicidal ideation as determined by a score of 2 points or higher on the Columbia Suicide Severity Rating Scale
5. suicidal behavior in the past 6 months
6. contraindication to recombinant human growth hormone (rhGH) such as hypersensitivity to rhGH or any of the components of the supplied product
7. acute medical illness, active infection, cancer, or decompensated chronic medical illness (e.g., decompensated diabetes mellitus, congestive heart failure, chronic obstructive pulmonary disease)
8. evidence of substance use disorder in the past 6 months other than mild alcohol or cannabis use disorder diagnosed by clinician at time of screening.
9. urine toxicology evidence of illicit drug use (excluding cannabis) within the past 90 days prior to screening
10. BMI > 35 or body weight > 350 lbs
11. abnormal pituitary anatomy documented by an MRI using a Sella protocol
12. women who are pregnant or of child-bearing potential who are unable/unwilling to use one of the following barrier contraceptives: condoms, diaphragm, cervical cap, or intrauterine device
13. current use of the following: growth hormone, estrogen or estrogen-like dietary supplements, hormonal contraceptives, progestin, insulin growth factor 1 (IGF-1), or chronic glucocorticoid use in supraphysiologic doses

15) currently enrolled in any other interventional drug trials unless prior approval is provided by the study chairs and the study sponsor

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in truncal fat mass from baseline to six months | 6 months
  The primary outcome measure is the difference of truncal fat mass percentage from baseline to six months. Truncal fat mass will be assessed at baseline, 3-months, and 6-months using calibrated dual energy x-ray absorptiometry (DEXA). A large mean difference corresponds with greater changes in truncal fat mass. Decreased truncal fat mass is associated with reduced risk of cardiovascular disease.

SECONDARY OUTCOMES:
Cardiometabolic Risk Factors | 6 months
  Change in cardiometabolic risk factors from baseline to 6 months measured by fasting low density lipoproteins (LDL) and highly sensitive C-reactive protein levels. A decrease in lipoprotein corresponds with increased lipoprotein metabolism, and lower C-reactive protein levels corresponds with less inflammation. A reduction in both suggests lower risk of cardiometabolic disease.
Lean body mass | 6 months
  The change in appendicular lean body mass between baseline and 6 months will be assessed using calibrated dual energy x-ray absorptiometry. The difference will capture changes in body composition (fat and muscle) with a higher difference corresponding with greater body composition changes.
Assessment of quality of life | 6 months
  Change in the quality of life from baseline to 6 months will be measured by the Quality of Life questionnaire for Adult Growth Hormone Deficiency. The score ranges from 0 to 25, with a score of 25 representing highest symptomatic burden and lower quality of life. A change in score is positively correlated with the patient's perception of treatment benefit, and a score change of 3.5 points is considered clinically meaningful.
Fatigue | 6 months
  Fatigue will be measured using the Fatigue Severity Scale. The questionnaire minimum score is a 9 and maximum score is 63. Higher scores represent greater fatigue severity.
Depression, Anxiety, and Stress | 6 months
  The Depression, Anxiety, and Stress Scale-21 (DASS-21), a 21-item questionnaire, will be used to assess depression, anxiety, and stress symptoms. The score range is 0 - 126 with a higher score representing greater severity or frequency of negative emotional symptoms.
Pain Intensity and Interference | 6 months
  Pain intensity and interference will be assessed using the Defense and Veterans Pain Rating Scale. The questionnaire contains two sections, one assessing current level of pain and the other evaluating the extent to which pain interferes with biopsychosocial factors such as daily activity, sleep, mood, and stress. The minimum score for each section is 0 and maximum score is 10 where higher scores correspond with more intense pain and greater interference.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Jorge, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Michael E. DeBakey VA Medical Center, Houston, Texas
  - VA Puget Sound Healthcare System, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The data supporting the findings in this study may be made available upon request to VA and non-VA researchers in accordance to VA policy.
Time Frame: Data will be available up to 24 months after article publication.
Access Criteria: Access to trial data can be requested by qualified researchers engaging in independent scientific research and will be provided following the review and approval of a research proposal, statistical analysis plan, and data usage agreement.